CLINICAL TRIAL: NCT00775684
Title: A Randomized, Controlled Trial Comparing the Effect of Exenatide, Sitagliptin or Glimepiride on Functional ß -Cell Mass in Patients With Impaired Fasting Glucose or Early Type 2 Diabetes
Brief Title: Effect of Exenatide, Sitagliptin or Glimepiride on Functional ß -Cell Mass
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Pennsylvania (Other)
Collaborators: Pennsylvania Department of Health (Other Government)
Responsible Party: Principal Investigator, Michael R. Rickels, MD, MS, Professor of Medicine, University of Pennsylvania
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 808425
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Results first posted 2017-12-06 (Actual); Last update posted 2022-06-07 (Actual); Status verified 2022-05

CONDITIONS: Pre-diabetes; Type 2 Diabetes
Keywords: Exenatide; Sitagliptin; Glimepiride; Glucagon-Like Peptide-1; Impaired Fasting Glucose; Type 2 Diabetes; Beta-cell Function; Beta-cell Secretory Capacity; Glucose-potentiated arginine
MeSH Terms: conditions — Glucose Intolerance; Diabetes Mellitus, Type 2 | interventions — Exenatide; Sitagliptin Phosphate; glimepiride

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Exenatide (Experimental): Exenatide (Byetta®)-5 µg injected subcutaneously twice daily and increased after 1 month to 10 µg twice daily as tolerated by gastrointestinal effects
  Interventions: Drug: Exenatide
- Sitagliptin (Experimental): Sitagliptin (Januvia®)-100 mg by mouth every morning
  Interventions: Drug: Sitagliptin
- Glimepiride (Active Comparator): Glimepiride (Amaryl®)-0.5 mg by mouth every morning and then increased by 0.5 - 1.0 mg at each monthly visit to achieve an average fasting glucose < 110mg/dl
  Interventions: Drug: Glimepiride

INTERVENTIONS:
Drug: Exenatide — Exenatide (Byetta®)-5 µg injected subcutaneously twice daily and increased after 1 month to 10 µg twice daily as tolerated by gastrointestinal effects
  Other Names: Byetta®
  Arms: Exenatide
Drug: Sitagliptin — Sitagliptin (Januvia®)100 mg by mouth every morning
  Other Names: Januvia®
  Arms: Sitagliptin
Drug: Glimepiride — Glimepiride (Amaryl®)-0.5 mg by mouth every morning and then increased by 0.5 - 1.0 mg at each monthly visit to achieve an average fasting glucose < 110mg/dl
  Other Names: Amaryl®
  Arms: Glimepiride

SUMMARY:
This study evaluates exenatide, sitagliptin, and glimepiride for the treatment of high blood sugar in patients with impaired fasting glucose or early type 2 diabetes. The purpose of this study is to determine if exenatide and sitagliptin increase the amount of insulin made by the pancreas compared to glimepiride. It is hypothesized that exenatide or sitagliptin will sustain or increase the amount of insulin made by the pancreas in comparison to glimepiride.

DETAILED DESCRIPTION:
The incidence of type 2 diabetes (T2D) has reached epidemic proportions throughout the world. In the United States more than 1.5 million new cases of diabetes were diagnosed in 2005, and the estimated prevalence of the disease was over 20 million. Another 54 million Americans are believed to have impaired fasting glucose, which represents a "pre-diabetic" state at increased risk for progression to overt diabetes. T2D ultimately results from an inadequate mass of functional beta-cells, where insufficient beta-cell compensation for insulin resistance leads to the development of impaired glucose tolerance and eventually diabetes. Autopsy studies have demonstrated a decreased beta-cell mass occurring with fasting glucose > 110 mg/dl, consistent with functional studies that demonstrate decreased beta-cell (insulin) secretory capacity beginning in the range of impaired fasting glucose. Strategies that might preserve or expand functional beta-cell mass in vivo would be expected to reverse the progressive deterioration in blood glucose control seen with diabetes. One such strategy involves the incretin hormone glucagon-like peptide-1 (GLP-1), which is trophic for islet beta-cells, having both pro-proliferative and anti-apoptotic effects. However, it is not known whether increasing GLP-1 effects can preserve or enhance functional beta-cell mass in humans. This proposal will determine the effect of increasing GLP-1 levels on functional beta-cell mass in human subjects with impaired fasting glucose (fasting glucose 110 - 126 mg/dl) or early T2D (fasting glucose 127 - 149 mg/dl) where a critical window exists for reversing further beta-cell deterioration. GLP-1 effects will be promoted by administration of either the GLP-1 analog, exenatide, or by increasing endogenous GLP-1 levels through administration of the oral dipeptidyl peptidase 4 (DPP4) inhibitor sitagliptin for a 6-month period. To control for the effect of exenatide and sitagliptin on normalization of blood glucose, subjects will be randomized to receive exenatide, sitagliptin or the sulfonylurea glimepiride, the latter being a first-line anti-diabetogenic agent that will serve as an active comparator.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients age 18 to 70 years.
2. Ability to provide written informed consent
3. Mentally stable and able to comply with the procedures of the study protocol
4. Clinical history compatible with impaired fasting glucose or early T2D as defined by a plasma glucose concentration between 110-159 mg/dl following a 12 hour overnight fast performed off any anti-diabetogenic agent for at least 2 weeks (6 weeks for thiazolidinediones)
5. Stable body weight (+ 5%) for at least 2 weeks
6. Female Patients: Agree to use adequate contraception if reproductively capable. Adequate contraception includes either a hormonal or barrier method, or surgical sterilization.

Exclusion Criteria:

1. Diagnosis of type 1 diabetes
2. Receiving insulin, exenatide (Byetta®), or sitagliptin (Januvia®) treatment or taking > 2 oral anti-diabetogenic agents for the treatment of diabetes
3. BMI > 44 kg/m2
4. Allergy to any sulfa-containing compounds
5. Uncontrolled hypertension (Systolic Blood Pressure >160 or Diastolic Blood Pressure > 100 mmHg)
6. Uncontrolled hyperlipidemia (triglycerides > 500 or LDL > 160 mg/dl)
7. Elevation of liver function tests > 2 times the upper limit of normal
8. Estimated Glomerular Filtration Rate (GFR) < 55 ml/min/1.73m2 (46)
9. Hyperkalemia (serum potassium > 5.5 mmol/L)
10. Moderate anemia (hemoglobin concentration < 12 g/dl in men and < 11 g/dl in women)
11. Female patients: pregnant or lactating
12. Hepatic cirrhosis
13. Known active alcohol or substance abuse
14. Active cardiovascular disease
15. Use of any investigational agent within 6 weeks of the baseline visit
16. Any medical condition that, in the opinion of the investigator, will interfere with the safe completion of the trial

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2008-10; Primary Completion 2012-11 (Actual); Study Completion 2012-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Rickels, M.D., M.S., Principal Investigator — University of Pennsylvania, Division of Endocrinology, Diabetes & Metabolism
Locations (3):
- United States (3):
  - Clinical and Translational Research Center, Hospital of University of Pennsylvania, Philadelphia, Pennsylvania
  - Rodebaugh Diabetes Center, Hospital of the University of Pennsylvania, Philadelphia, Pennsylvania
  - Pennsylvania Hospital, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] National Diabetes Statistics http://diabetes.niddk.nih.gov/dm/pubs/statistics/index.htm 2005. 2-16-2007 Ref Type: Electronic Citation
- [Background] King H, Aubert RE, Herman WH. Global burden of diabetes, 1995-2025: prevalence, numerical estimates, and projections. Diabetes Care. 1998 Sep;21(9):1414-31. doi: 10.2337/diacare.21.9.1414. PMID 9727886
- [Background] U.K. prospective diabetes study 16. Overview of 6 years' therapy of type II diabetes: a progressive disease. U.K. Prospective Diabetes Study Group. Diabetes. 1995 Nov;44(11):1249-58. PMID 7589820
- [Background] Butler AE, Janson J, Bonner-Weir S, Ritzel R, Rizza RA, Butler PC. Beta-cell deficit and increased beta-cell apoptosis in humans with type 2 diabetes. Diabetes. 2003 Jan;52(1):102-10. doi: 10.2337/diabetes.52.1.102. PMID 12502499
- [Background] Ritzel RA, Butler AE, Rizza RA, Veldhuis JD, Butler PC. Relationship between beta-cell mass and fasting blood glucose concentration in humans. Diabetes Care. 2006 Mar;29(3):717-8. doi: 10.2337/diacare.29.03.06.dc05-1538. No abstract available. PMID 16505537
- [Background] Kahn SE. Clinical review 135: The importance of beta-cell failure in the development and progression of type 2 diabetes. J Clin Endocrinol Metab. 2001 Sep;86(9):4047-58. doi: 10.1210/jcem.86.9.7713. No abstract available. PMID 11549624
- [Background] Godsland IF, Jeffs JAR, Johnston DG. Loss of beta cell function as fasting glucose increases in the non-diabetic range. Diabetologia. 2004 Jul;47(7):1157-1166. doi: 10.1007/s00125-004-1454-z. Epub 2004 Jul 13. PMID 15249997
- [Background] Ward WK, Bolgiano DC, McKnight B, Halter JB, Porte D Jr. Diminished B cell secretory capacity in patients with noninsulin-dependent diabetes mellitus. J Clin Invest. 1984 Oct;74(4):1318-28. doi: 10.1172/JCI111542. PMID 6384269
- See also: Michael R. Rickels, M.D., M.S. Faculty Bio — http://www.med.upenn.edu/apps/faculty/index.php/g343/p32032
- See also: Rodebaugh Diabetes Center — http://pennhealth.com/diabetes/hup/
- See also: Center for Human Phenomic Science (Formerly the Clinical and Translational Research Center) — http://www.itmat.upenn.edu/chps/
- See also: Institute for Diabetes, Obesity & Metabolism - Clinical Trials — http://www.med.upenn.edu/idom/trials_rickels-bcell.html

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment is now closed for this study. All subject follow-up was completed in the spring of 2012.
  The purpose of the study was to evaluate three medications for the treatment of high blood sugar.
Period: Overall Study
Arm/Group | Exenatide | Sitagliptin | Glimepiride
Started | 17 | 13 | 17
Completed | 14 | 12 | 14
Not Completed | 3 | 1 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Exenatide | Sitagliptin | Glimepiride | Total
Number analyzed (Participants) | 17 | 13 | 17 | 47
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 17 | 13 | 17 | 47
  >=65 years | 0 | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 57 (2) | 57 (3) | 52 (3) | 55.3 (2.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 7 | 17
  Male | 11 | 9 | 10 | 30
Region of Enrollment [Number; unit: participants]
  United States | 17 | 13 | 17 | 47

OUTCOME MEASURES:

1. Primary Outcome: Effect on Functional Beta-cell Mass as Determined by Change in ß-cell Secretory Capacity at 6 Months (μU/ml)
Description: The acute insulin response to arginine (AIRarg) performed during the 340mg/dl glucose clamp allows for estimation of the the beta-cell secretory capacity (AIRmax) or functional beta-cell mass. Changes from baseline to 6 months of AIRmax were compared across groups
Time Frame: Baseline and 6 months
Population: We conducted a randomized controlled trial in 40 adult subjects with early Type 2 diabetes (T2D) who received the
  glucagon-like peptide (GLP-1) analog exenatide, the dipeptidyl peptidase IV inhibitor sitagliptin or the sulfonylurea glimepiride as an active comparator insulin secretagogue for 6 months.
Measure: Mean (Standard Error); unit: μU/ml
Arm/Group | Exenatide | Sitagliptin | Glimepiride
Number analyzed (Participants) | 14 | 12 | 14
μU/ml
  Acute Insulin Response (AIRmax)Baseline | 214 (60) | 149 (20) | 133 (19)
  Acute Insulin Response (AIRmax) 6 Months | 188.5 (34.6) | 158.3 (30.3) | 202.5 (35.1)
Statistical Analysis 1: Comparison: Exenatide vs Glimepiride; Student t test; Test type: Superiority; p = 0.1, t-test, 2 sided
Statistical Analysis 2: Comparison: Glimepiride; Repeated measure (baseline and 6 months); Test type: Superiority; p < 0.05, t-test, 2 sided

2. Secondary Outcome: Change in Acute Insulin Response to Arginine. (AIRarg)
Description: The changes in B-cell insulin secretion, Acute Insulin Response to arginine (AIRarg) after 6 months were compared to baseline AIRarg for each group. Listed below are AIRarg at baseline and 6 months for each group.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: uU/mL
Groups:
- AIRarg Exenatide; AIRarg Sitagliptin; AIRarg Glimepiride: Acute insulin response to arginine
Arm/Group | AIRarg Exenatide | AIRarg Sitagliptin | AIRarg Glimepiride
Number analyzed (Participants) | 14 | 12 | 14
uU/mL
  Acute Insulin Response (AIRarg) Baseline | 52 (14) | 35 (4) | 44 (6)
  Acute Insulin Response (AIRarg) 6 Months | 52 (11) | 34 (6) | 42 (4)
Statistical Analysis 1: Comparison: AIRarg Exenatide vs AIRarg Glimepiride; Within group changes over 6 months (delta= final - baseline) were compared; Test type: Superiority; p > 0.1, t-test, 1 sided

3. Secondary Outcome: Insulin Sensitivity at Baseline and 6 Months
Description: Insulin sensitivity (M/I) was determined by dividing the mean glucose infusion rate required during the 230 mg/dL glucose clamp (M) by the mean prestimulus insulin level (I) between 40 and 45 min of the glucose infusion The mean difference after 6 months in insulin sensitivity (M/I) were compared
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: ((mg/kg) /min) /uU/mL
Groups:
- M/I Exenatide; M/I Sitagliptin; M/I Glimepiride: Change in insulin sensitivity
Arm/Group | M/I Exenatide | M/I Sitagliptin | M/I Glimepiride
Number analyzed (Participants) | 14 | 12 | 14
((mg/kg) /min) /uU/mL
  M/I Baseline | 0.3 (0.1) | 0.3 (0.0) | 0.3 (0.1)
  M/I 6 Months | 0.3 (0.1) | 0.3 (0.1) | 0.3 (0.1)
Statistical Analysis 1: Comparison: M/I Exenatide vs M/I Sitagliptin vs M/I Glimepiride; To determine if exenatide or sitagliptin induced significant changes from baseline, the change for each measure (Δ = final - baseline) for each group was compared with the change in the glimepiride group using independent Student t tests; Test type: Superiority; p > 0.1, t-test, 1 sided

4. Secondary Outcome: PG 50 (the Plasma Glucose Level at Which Half-maximal Insulin Secretion is Achieved During the Glucose-potentiated Arginine Test) at Baseline and 6 Months
Description: Between ∼60 and 250 mg/dL, the magnitude of AIRarg is a linear function of the plasma glucose level, so the difference in AIRarg at fasting and 230 mg/dL glucose levels divided by the difference in plasma glucose (ΔAIRarg/ΔPG) gives the glucose-potentiation slope (GPS) (8,24-26). Using the y-intercept (b) from the line created by these two points, the plasma glucose level at which half-maximal insulin secretion is achieved (PG50) is derived from solving the equation 1/2 (AIRmax) = (GPS · PG50) + b, and provides a measure of β-cell sensitivity to glucose The mean difference after 6 months in PG 50 were compared. Listed below are the PG50 values at baseline and 6 months.
Time Frame: Baseline and 6 months
Measure: Mean (Standard Error); unit: mg/dL
Groups:
- P50 Exenatide; P50 Sitagliptin; P50 Glimepiride: Plasma glucose level at which half-maximal insulin secretion is achieved during the glucose-potentiated arginine test
Arm/Group | P50 Exenatide | P50 Sitagliptin | P50 Glimepiride
Number analyzed (Participants) | 14 | 12 | 14
mg/dL
  PG50 Baseline | 175 (13) | 226 (12) | 168 (17)
  PG50 6 Months | 190 (14) | 209 (16) | 182 (10)
Statistical Analysis 1: Comparison: P50 Exenatide vs P50 Sitagliptin vs P50 Glimepiride; Test type: Superiority; p > 0.1, t-test, 1 sided

5. Primary Outcome: Effect on Functional Beta-cell Mass as Determined by Change in ß-cell Secretory Capacity at 6 Months (pg/mL)
Description: AGRmin is performed during the 340mg/dl glucose clamp allows for estimation of the minimum alpha-cell glucagon secretion. Changes from baseline to 6 months of AGRmin were compared across groups.
Time Frame: Baseline and 6 months
Population: as for outcome 1
Measure: Mean (Standard Error); unit: pg/mL
Arm/Group | Exenatide | Sitagliptin | Glimepiride
Number analyzed (Participants) | 14 | 12 | 14
pg/mL
  Acute Glucose Response (AGRmin) Baseline | 51 (12) | 55 (8) | 37 (6)
  Acute Glucose Response (AGRmin) 6 Months | 52 (12) | 59 (19) | 59 (8)

ADVERSE EVENTS:
Arm/Group | Exenatide | Sitagliptin | Glimepiride
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/13 | 0/17
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/13 | 0/17
Other Adverse Events (participants affected / at risk) | 0/17 | 0/13 | 0/17

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No